CLINICAL TRIAL: NCT00000243
Title: Transitioning Patients From Methadone to Buprenorphine/Naloxone for Treating Opioid Dependence
Brief Title: Effects of Buprenorphine/Naloxone in Treating Opioid Dependent Individuals Who Are Maintained on Methadone
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIDA-08045-1; R01-08045-1; DPMC
Record Dates: First submitted 1999-09-20; First posted 1999-09-21 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Opioid-Related Disorders
Keywords: opioid dependence
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Buprenorphine

INTERVENTIONS:
Drug: Buprenorphine

SUMMARY:
Buprenorphine is a drug that may be helpful in treating opioid dependent individuals who were previously maintained on methadone. The purpose of this study is to determine the effects of different doses of buprenorphine/naloxone in treating opioid dependent individuals who were previously maintained on methadone.

DETAILED DESCRIPTION:
Buprenorphine is a mixed agonist-antagonist opioid that is being developed as a treatment for opioid dependence. Because buprenorphine is a partial mu agonist opioid, under certain conditions it is possible for buprenorphine to precipitate opioid withdrawal in opioid dependent individuals. A person with a high level of physical dependence could experience buprenorphine-related precipitated withdrawal. The purpose of this study is to test the acute effects of different doses of buprenorphine/naloxone in opioid dependent individuals maintained on methadone. The study is designed to provide dosing schedules similar to those that might be initially used in a physician's office.

ELIGIBILITY:
Inclusion Criteria:

* Meets criteria for opioid dependence

Exclusion Criteria:

* Significant medical or psychiatric illness

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16
Dates: Start 2002-09; Study Completion 2004-01

PRIMARY OUTCOMES:
Physiological effects
Analog rating scale for drug effects

CONTACTS AND LOCATIONS:
Overall Officials: Eric C. Strain, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University (BPRU) Bayview Campus, Baltimore, Maryland, United States